CLINICAL TRIAL: NCT00375024
Title: Patient Navigator Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-14718
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer; Colon Cancer
Keywords: Patient navigation; Breast cancer; Colon cancer; Questionnaire
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Patient Navigator (Other): Patients will meet with a Patient Navigator regarding their treatment and any related concerns.
  Interventions: Procedure: Patient Navigation
- 2: Without Navigator (Other): Patient will work with existing clinic staff, which does not include a Patient Navigator.
  Interventions: Procedure: Clinic Staff

INTERVENTIONS:
Procedure: Patient Navigation — Inclusion of Patient Navigator in treatment plan.
  Arms: 1: Patient Navigator
Procedure: Clinic Staff — Specific Patient Navigator will not be included in treatment plan. Existing clinical staff will work with the patients.
  Arms: 2: Without Navigator

SUMMARY:
Patient Navigation is a Supportive Care Intervention that addresses barriers to quality standard care by providing individualized assistance to patients and families. The NCI is conducting several research programs to test the effectiveness of this approach. The expected outcomes of patient navigation through the cancer care system include:

* Timely, definitive diagnosis following an abnormal test
* Timely treatment following positive diagnosis
* Patient satisfaction with the diagnostic and care system experience

DETAILED DESCRIPTION:
The goal of our local project is to provide Tampa Bay with a culturally appropriate Patient Navigator Program that will decrease delay in diagnosis and delivery of cancer care in an acceptable and cost-effective manner leading to lower cancer mortality among our underserved populations. We will partner with community health centers in the Tampa Bay area to provide an avenue for patients who have received an abnormal screening for breast and colorectal cancer to easier pilot the course of the healthcare system. The populations served by this program will include African-Americans, Hispanics and rural Whites who are medically underserved due to lack of insurance, documentation issues and a variety of other barriers to health care.

The primary outcome to be tested with this program is the time it takes for patients with an abnormality to receive a definitive diagnosis. Secondary outcomes such as patient satisfaction and cost-effectiveness will also be measured. This program occurs in three phases. In Phase I, the aim is to work closely with our key community partners to conduct formative research for the development of an acceptable, appealing, and appropriate Patient Navigator Program. The aim for Phase II is to conduct a group randomized controlled trial by having participating clinics randomly assigned to an intervention or control clinic. The outcomes from this phase in the project will be assessed through chart reviews, patient satisfaction surveys and other survey methods. In Phase III a comprehensive evaluation on the program will be produced and disseminated nationally.

ELIGIBILITY:
Inclusion Criteria:

* Receive health care at one of the enrolled clinics
* Newly diagnosed with breast of colorectal cancer or if they have an abnormality that is suspicious for breast (breast lump, or abnormal mammogram) or colorectal cancer (abnormal colon screening test, blood in bowel movement).

Exclusion Criteria:

* Persons with previous history of breast or colon cancer will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1267 (Actual)
Dates: Start 2007-05; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Questionnaire Results Regarding Time to Diagnosis | Individual per patient
  Time from finding of abnormality to definitive diagnosis

SECONDARY OUTCOMES:
Patient Satisfaction Questionaire Results | At end of patient participation
Questionnaire Results Regarding Patient Navigators | End of study
  To determine if patient navigators are cost effective

CONTACTS AND LOCATIONS:
Overall Officials: Richard Roetzheim, MD, MSPH, Principal Investigator — University of South Florida
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Battaglia TA, Darnell JS, Ko N, Snyder F, Paskett ED, Wells KJ, Whitley EM, Griggs JJ, Karnad A, Young H, Warren-Mears V, Simon MA, Calhoun E. The impact of patient navigation on the delivery of diagnostic breast cancer care in the National Patient Navigation Research Program: a prospective meta-analysis. Breast Cancer Res Treat. 2016 Aug;158(3):523-34. doi: 10.1007/s10549-016-3887-8. Epub 2016 Jul 18. PMID 27432417
- [Derived] Wells KJ, Winters PC, Jean-Pierre P, Warren-Mears V, Post D, Van Duyn MA, Fiscella K, Darnell J, Freund KM; Patient Navigation Research Program Investigators. Effect of patient navigation on satisfaction with cancer-related care. Support Care Cancer. 2016 Apr;24(4):1729-53. doi: 10.1007/s00520-015-2946-8. Epub 2015 Oct 5. PMID 26438146
- [Derived] Rodday AM, Parsons SK, Snyder F, Simon MA, Llanos AA, Warren-Mears V, Dudley D, Lee JH, Patierno SR, Markossian TW, Sanders M, Whitley EM, Freund KM. Impact of patient navigation in eliminating economic disparities in cancer care. Cancer. 2015 Nov 15;121(22):4025-34. doi: 10.1002/cncr.29612. Epub 2015 Sep 8. PMID 26348120
- [Derived] Ko NY, Darnell JS, Calhoun E, Freund KM, Wells KJ, Shapiro CL, Dudley DJ, Patierno SR, Fiscella K, Raich P, Battaglia TA. Can patient navigation improve receipt of recommended breast cancer care? Evidence from the National Patient Navigation Research Program. J Clin Oncol. 2014 Sep 1;32(25):2758-64. doi: 10.1200/JCO.2013.53.6037. Epub 2014 Jul 28. PMID 25071111
- [Derived] Lee JH, Fulp W, Wells KJ, Meade CD, Calcano E, Roetzheim R. Patient navigation and time to diagnostic resolution: results for a cluster randomized trial evaluating the efficacy of patient navigation among patients with breast cancer screening abnormalities, Tampa, FL. PLoS One. 2013 Sep 16;8(9):e74542. doi: 10.1371/journal.pone.0074542. eCollection 2013. PMID 24066145
- See also: H Lee Moffiitt Cancer Center & Research Institute website — http://www.moffitt.org